CLINICAL TRIAL: NCT01030705
Title: Common Sensing and Right Ventricular Automatic Capture
Brief Title: Common Sensing and Right Ventricular Automatic Capture (COGNATE)
Acronym: COGNATE
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: COGNATE
Record Dates: First submitted 2009-12-09; First posted 2009-12-11 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2011-09

CONDITIONS: Bradycardia; Chronotropic Incompetence
Keywords: Bradycardia; pacemaker
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will collect data on features for future pacemakers via an external non-implantable system.

DETAILED DESCRIPTION:
COGNATE is an acute, confirmatory prospective, multi-center study designed to gather data on Brady and CRT-P indicated patients, with no restrictions on the type/brand of leads. This study will enroll up to 80 patients in up to 12 centers. Total duration of the study is expected to be 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to receive either Pacemaker (dual chamber) or CRT-P devices based on physician discretion
* Patients who are willing and capable of participating in all testing associated with this Clinical Investigation
* Patients who are age 18 or above, or of legal age to give informed consent specific to state and national law

Exclusion Criteria:

* Patient enrolled in any concurrent study, without Boston Scientific CRM written approval, that may confound the results of this study
* Patients with a prosthetic mechanical tricuspid heart valve
* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir Saba, MD, Principal Investigator — Health Care Conusltant
Locations (5):
- United States (5):
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Nebraska Heart Institute, Lincoln, Nebraska
  - University of Pittsburgh Medical Center, Cardiac Electrophysiology, Pittsburgh, Pennsylvania
  - Intermountain Medical Center, Murray, Utah
  - Virginia Commonwealth University Health System, Medical College of Virginia, MCV Physicians and Hospitals, Richmond, Virginia